CLINICAL TRIAL: NCT06313190
Title: Stereotactic Body Radiotherapy with or Without Adjuvant Immunotherapy for Small Hepatocellular Carcinoma: an Open-label, Randomized, Phase II Trial
Brief Title: Combination of SBRT and Immunotherapy in Small Hepatocellular Carcinoma (HSBRT2402)
Acronym: HSBRT2402
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Ningbo Medical Center Lihuili Eastern Hospital (Unknown)
Responsible Party: Principal Investigator, Mian XI, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2024-061
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Immunotherapy; Stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Patients in both cohorts will receive SBRT using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3 fractions over 1 week. Then patients in the study group (arm A) will receive sintilimab as adjuvant therapy for up to 6 cycles after the completion of radiotherapy.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Sintilimab
- Arm B (Active Comparator): Patients in both cohorts will receive SBRT using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3 fractions over 1 week. Then patients in the control group (arm B) will be followed up regularly.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Patients in both cohorts will receive SBRT using volumetric arc therapy. The prescribed dose is 30-54 Gy in 3 fractions over 1 week.
  Other Names: SBRT
Drug: Sintilimab — Patients received sintilimab 200 mg every 3 weeks for up to 6 cycles, with the first dose within 1 week after the completion of SBRT.
  Other Names: IBI308
  Arms: Arm A

SUMMARY:
For inoperable small hepatocellular carcinoma (HCC), stereotactic body radiotherapy (SBRT) is an effective and safe local treatment. Despite satisfactory local control rate, the incidence of recurrence out the field remains substantial, with 2-year PFS of 31.9% to 60.9%. Therefore, a more effective treatment mode is urgently needed. Immune checkpoint inhibitors targeting PD-1/PD-L1 have shown substantial clinical benefits in advanced HCC as well as resected high-risk HCC. Recently, the combination of immunotherapy with SBRT has shown promising activity in HCC, but its utility in small HCC is unclear. The aim of this study was to investigate the efficacy and safety of SBRT followed by sintilimab (an anti-PD-1 antibody) in patients with recurrent or residual small HCC.

DETAILED DESCRIPTION:
A total of 140 patients with recurrent or residual small HCC will be stratified according to tumor diameter (≤3 vs. >3 cm) and tumor type (recurrent vs. residual) and randomly assigned (1:1) to receive stereotactic body radiotherapy (SBRT) with or without adjuvant sintilimab for 6 cycles (200 mg, once every 3 weeks, with the first dose within 1 week after the completion of SBRT).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed hepatocellular carcinoma or diagnosed by American Association for the Study of Liver Disease criteria;
2. Presence of recurrent or residual HCC lesions without vascular invasion or extrahepatic metastasis confirmed by CT or MRI, the sum of the maximum diameter of lesions ≤5 cm, total number of lesions were ≤2, and at least one of which is measurable according to the RECIST 1.1 Criteria;
3. Previous molecular targeted therapy or intravenous chemotherapy is allowed, but the interval of drug withdrawal was at least 6 months prior to protocol therapy;
4. Age at diagnosis 18 to 75 years;
5. Eastern Cooperative Oncology Group performance status ≤ 2
6. Child-Pugh class A liver function;
7. Normal liver volume greater than 700 ml;
8. Estimated life expectancy ≥24 weeks;
9. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 3.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 50×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
10. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have previously been treated with immune checkpoint inhibitors;
2. Patients with extrahepatic metastasis disease;
3. A history of abdominal radiotherapy;
4. Known or suspected allergy or hypersensitivity to monoclonal antibodies;
5. Patients who have a preexisting or coexisting bleeding disorder;
6. Female patients who are pregnant or lactating;
7. Inability to provide informed consent due to psychological, familial, social and other factors;
8. A history of malignancies other than hepatocellular carcinoma before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer;
9. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
10. Patients who cannot tolerate radiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia;
11. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
12. A history of interstitial lung disease or non-infectious pneumonia;
13. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
15. Any unstable situation that may endanger the safety and compliance of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | From date of enrollment until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months
  Two-year follow-up from the date of enrollment to the date of disease progression or last follow-up

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 36 months
  Three-year follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Local control rate (DCR) | From date of enrollment to the date of last follow-up, assessed up to 36 months
  The proportion of patients with complete response, partial response, or stable disease for the target lesion according to RECIST criteria.
Treatment-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0.

OTHER OUTCOMES:
Correlation between serum cytokines and overall survival and immune-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months
  The correlation between dynamic change of serum cytokines (IL-2R, IL-6, IL-13, IL-8, CCL3, CD40, and CD274) during treatment and survival outcomes and immune-related adverse events.
Correlation between ctDNA and overall survival | From date of enrollment to the date of last follow-up, assessed up to 36 months
  The correlation between dynamic change of ctDNA (before and after treatment) and survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Kim HJ, Park S, Kim KJ, Seong J. Clinical significance of soluble programmed cell death ligand-1 (sPD-L1) in hepatocellular carcinoma patients treated with radiotherapy. Radiother Oncol. 2018 Oct;129(1):130-135. doi: 10.1016/j.radonc.2017.11.027. Epub 2018 Jan 30. PMID 29366520
- [Background] Chiang CL, Chiu KWH, Chan KSK, Lee FAS, Li JCB, Wan CWS, Dai WC, Lam TC, Chen W, Wong NSM, Cheung ALY, Lee VWY, Lau VWH, El Helali A, Man K, Kong FMS, Lo CM, Chan AC. Sequential transarterial chemoembolisation and stereotactic body radiotherapy followed by immunotherapy as conversion therapy for patients with locally advanced, unresectable hepatocellular carcinoma (START-FIT): a single-arm, phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):169-178. doi: 10.1016/S2468-1253(22)00339-9. Epub 2022 Dec 15. PMID 36529152
- [Background] Wang K, Xiang YJ, Yu HM, Cheng YQ, Liu ZH, Qin YY, Shi J, Guo WX, Lu CD, Zheng YX, Zhou FG, Yan ML, Zhou HK, Liang C, Zhang F, Wei WJ, Lau WY, Li JJ, Liu YF, Cheng SQ. Adjuvant sintilimab in resected high-risk hepatocellular carcinoma: a randomized, controlled, phase 2 trial. Nat Med. 2024 Mar;30(3):708-715. doi: 10.1038/s41591-023-02786-7. Epub 2024 Jan 19. PMID 38242982
- [Background] Ren Z, Xu J, Bai Y, Xu A, Cang S, Du C, Li Q, Lu Y, Chen Y, Guo Y, Chen Z, Liu B, Jia W, Wu J, Wang J, Shao G, Zhang B, Shan Y, Meng Z, Wu J, Gu S, Yang W, Liu C, Shi X, Gao Z, Yin T, Cui J, Huang M, Xing B, Mao Y, Teng G, Qin Y, Wang J, Xia F, Yin G, Yang Y, Chen M, Wang Y, Zhou H, Fan J; ORIENT-32 study group. Sintilimab plus a bevacizumab biosimilar (IBI305) versus sorafenib in unresectable hepatocellular carcinoma (ORIENT-32): a randomised, open-label, phase 2-3 study. Lancet Oncol. 2021 Jul;22(7):977-990. doi: 10.1016/S1470-2045(21)00252-7. Epub 2021 Jun 15. PMID 34143971